CLINICAL TRIAL: NCT02876211
Title: Benefits of the Paricalcitol (Selective Vitamin D Receptor Activator) on Anemia of Inflammation in Dialysis Patients Under Erythropoiesis-stimulating Agents Treatment.
Brief Title: Paricalcitol Improves Anemia of Inflammation
Acronym: PIERAID
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficult inclusion of patients diagnosed with renal anemia in chronic hemodialysis patients without hyperparathyroidism.
Sponsor: Hospital Son Espases (Other)
Responsible Party: Principal Investigator, Miguel Giovanni Uriol Rivera, Ph.D. MD., Hospital Son Espases
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PIERAID-2013
Record Dates: First submitted 2016-08-12; First posted 2016-08-23 (Estimated); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Anemia
Keywords: Renal disease; Erythropoiesis; Erythropoietin stimulating agent; Iron; Klotho; Selective vitamin D receptor activation
MeSH Terms: conditions — Anemia; Kidney Diseases | interventions — paricalcitol; epoetin beta

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- paricalcitol plus epoetin beta (Experimental): Paricalcitol 2 capsules /three times per week & epoetin
  Interventions: Drug: Paricalcitol; Drug: Epoetin beta
- placebo plus epoetin beta (Placebo Comparator): Placebo 2 capsules/three times per week & epoetin
  Interventions: Drug: Epoetin beta; Drug: Placebo

INTERVENTIONS:
Drug: Paricalcitol — Paricalcitol 2 capsules/three times per week
  Other Names: Selective vitamin D receptor activation
  Arms: paricalcitol plus epoetin beta
Drug: Epoetin beta — epoetin 1-3 times per week
  Other Names: anti-anemic drug
Drug: Placebo — Placebo 2 capsules/three times per week
  Arms: placebo plus epoetin beta

SUMMARY:
Anemia of inflammation (AI) is a common comorbidity in hemodialysis patients. Paricalcitol is a selective vitamin D receptor activator with potential benefits on anti-inflammatory cytokines expression. The paricalcitol for the secondary hyperparathyroidism control may improve AI decreasing erythropoietin stimulating agents (ESAs) dosage.

DETAILED DESCRIPTION:
Anemia of inflammation and secondary hyperparathyroidism (SHPT) are two common clinical complications in patients with chronic kidney disease. Eryptosis (accelerated red blood cell death) is a novel mechanism associated with renal anemia and several factors such us iron, erythropoietin and klotho (anti-aging hormone) deficiency have been associated with this process.

The use of the paricalcitol may inhibit pro-inflammatory cytokines expression, especially interleukine-6, which is one of the most important cytokine associated with the pathogenesis of the AI. If the use of the paricalcitol for the SHPT control may exert direct influence on the erythropoiesis process is not known.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years.
* Patients with CKD on hemodialysis of any etiology..
* Hemoglobin between 9 and 12g/dl at least 12 weeks before enrollment in the study.
* Hemoglobin plasma levels stabilized: Hb variation <or = 1 g / dl for the two months prior to inclusion in the study.
* Patients with anemia of renal etiology.
* ESA treatment with stable doses for 2 months prior to baseline.Stable dose ESA Definition: Variation <or = 3000UI/week.
* Iron status: Ferritin> 200 ng / mL and/or transferrin saturation index (IST):> = 20%).
* KT / V >= 1.2 ( Daugirdas-2nd generation).
* Calcium concentrations between : 8.4 to 9.5 mg / dl and phosphorus: 3.5-5.5 mg / dl.
* Vitamin D 25OH normal >= 15 ng / ml (patients with lower levels will be supplemented with calcifediol 16000 IU / bi-weekly for 6 weeks in selected patients).
* PTHi concentrations> = 150 pg / mL and <or = to 300 pg / ml.
* Patients who accept their inclusion in the study and sign informed consent.

Exclusion Criteria:

* Epoetin beta dose > 18,000 IU / weekly.
* Pregnant woman of childbearing age or gestational wishes or not to use adequate contraception ( the Ogino-Knaus contraceptive method is considered unsuitable).
* Active bleeding episode or history of transfusion the 2 months prior to baseline.
* Patients with non-renal causes of anemia: malignancies, folic acid or vitamin B12 deficiency, hemoglobinopathies, hemolysis, pure red cell aplasia secondary to erythropoietin.
* Patients treated with the selective vitamin D receptor activator in the 3 months prior to inclusion in the study.
* Acute or chronic symptomatic: heart failure (IV-NYHA), infection or inflammatory disease, uncontrolled hypertension that requires the suspension of epoetin beta, thrombocytopathies, aplastic anemia.
* Immunosuppressive treatment with uncontrolled Hemoglobin level
* Allergy to paricalcitol or any of its components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2022-08 (Actual); Study Completion 2024-12 (Actual)

PRIMARY OUTCOMES:
Changes in ESA dosage | 6 months
  Percentage of ESA doses after 6 months of the paricalcitol or placebo administration.

SECONDARY OUTCOMES:
Changes on ferrokinetics. | 6 months
  Changes on serum iron, transferrin, ferritin, transferrin saturation and red cell distribution width at month 6.
Changes on interleukin-6 plasma levels. | 6 months
  Changes on pg/ml
Changes on hepcidin plasma levels. | 6 months
  Changes on pg/ml
Changes on erythropoietin plasma levels. | 6 months
  Changes on mUI/ml
Changes on systolic blood pressure. | 6 months
  Changes in mmHg determined by 24 hours ambulatory blood pressure monitoring.
Changes on diastolic blood pressure. | 6 months
  Changes in mmHg determined by 24 hours ambulatory blood pressure monitoring.
Cardiovascular serious adverse events in each arm of treatment. | 6 months
  Cardiac arrest, angina pectoris. Stroke.
Adverse events related to vascular access disfunction. | 6 month
  Arteriovenous fistula site hemorrhage or thrombosis. Catheter disfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Uriol, Ph.D.M.D., Principal Investigator — Son Espases University Hospital
Locations (1):
- Son Espases University Hospital, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: Yes
The IPD could be shared with any interested public research institute
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After finalized the study
Access Criteria: Research

REFERENCES:
- [Background] Sun CC, Vaja V, Babitt JL, Lin HY. Targeting the hepcidin-ferroportin axis to develop new treatment strategies for anemia of chronic disease and anemia of inflammation. Am J Hematol. 2012 Apr;87(4):392-400. doi: 10.1002/ajh.23110. Epub 2012 Jan 31. PMID 22290531
- [Background] Perlstein TS, Pande R, Berliner N, Vanasse GJ. Prevalence of 25-hydroxyvitamin D deficiency in subgroups of elderly persons with anemia: association with anemia of inflammation. Blood. 2011 Mar 10;117(10):2800-6. doi: 10.1182/blood-2010-09-309708. Epub 2011 Jan 14. PMID 21239700
- [Background] Kempe DS, Ackermann TF, Fischer SS, Koka S, Boini KM, Mahmud H, Foller M, Rosenblatt KP, Kuro-O M, Lang F. Accelerated suicidal erythrocyte death in Klotho-deficient mice. Pflugers Arch. 2009 Jul;458(3):503-12. doi: 10.1007/s00424-009-0636-4. Epub 2009 Jan 28. PMID 19184092